CLINICAL TRIAL: NCT02617888
Title: The HEART BREAK Study: Effects of Heart Imaging Radiation on DNA Double-Stranded Breaks in Blood Lymphocytes and Hair Follicle Cells
Brief Title: Effects of Heart Imaging Radiation on DNA Double-Stranded Breaks in Blood Lymphocytes and Hair Follicle Cells
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Todd C. Villines, Director of Cardiovascular Research, Walter Reed National Military Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 362425
Record Dates: First submitted 2015-11-19; First posted 2015-12-01 (Estimated); Results first posted 2017-01-19 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Coronary Artery Disease; Chest Pain
Keywords: radiation; cardiac computed tomography; CCTA; breast shielding; Myocardial perfusion scintigraphy; MPS; Invasive coronary angiography; ICA
MeSH Terms: conditions — Coronary Artery Disease; Chest Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CCTA Breast Shields (Active Comparator): Within female subset, randomization to wearing bismuth breast shield.
  Interventions: Radiation: CCTA ~ BREAST SHIELDS
- CCTA No Breast Shields (No Intervention): Within female subset, randomization to wearing no bismuth breast shield (standard of care).
- Observational Arm (No Intervention): Non-females undergoing CTA and subjects undergoing cardiac catheterization and nuclear medicine testing.

INTERVENTIONS:
Radiation: CCTA ~ BREAST SHIELDS — Breast shield placement (randomized) among women.
  Other Names: BISMUTH BREAST SHIELDS
  Arms: CCTA Breast Shields

SUMMARY:
Purpose

1. To investigate the effects of cardiac imaging radiation on the induction of DNA double-strand breaks by enumerating gamma-H2AX foci in blood lymphocytes and plucked hair follicle cells.
2. To estimate whether the use of breast shields in cardiac computed tomographic angiography (CCTA) limits the effective radiation exposure of breast tissue.

DETAILED DESCRIPTION:
The primary objective of the study is to analyze blood and hair samples from patients undergoing cardiac imaging to estimate radiation exposure levels as well as their biological effects (i.e. to determine the degree of genotoxicity by measuring the amounts of DNA double-strand breaks).

The secondary objective is to investigate whether the use of in-plane breast shielding in female patients undergoing CT angiography (CCTA) limits the radiation exposure of breast tissue and subsequent DNA damage in blood lymphocytes and hair follicle cells.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female adult subjects (age greater than 18 years)
* Referred for cardiac computed tomography angiography (CCTA), myocardial perfusion scintigraphy (MPS), or diagnostic invasive coronary angiography (ICA).

Exclusion Criteria:

* Female patients that identify themselves as pregnant or have a positive pregnancy test prior to cardiac imaging.
* History (present or past) of leukemia or lymphoma.
* History of radiation therapy
* X-ray examination or scintigraphy within the last 72 hours.
* History of coronary revascularization (coronary artery bypass grafting or percutaneous coronary intervention)
* Patients undergoing percutaneous coronary intervention at completion of diagnostic left heart catheterization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2011-03; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd C Villines, MD, Principal Investigator — WRNMMC

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 101 patients enrolled in intervention arms (breast shields). Other patients in observational arm (not completed analysis).
Groups:
- CCTA Breast Shields: Within female subset, randomization to wearing bismuth breast shield.
  .
- CCTA No Breast Shields: Within female subset, randomization to not wearing bismuth breast shield (standard of care).
- Observational: Non-female patients undergoing coronary CTA, patients undergoing nuclear cardiology studies and invasive coronary angiography.
Period: Overall Study
Arm/Group | CCTA Breast Shields | CCTA No Breast Shields | Observational
Started | 50 | 51 | 127
Completed | 49 (Incomplete due to inadequate double-strand DNA break sample.) | 44 (Incomplete due to inadequate double-strand DNA break samples.) | 127
Not Completed | 1 | 7 | 0

BASELINE CHARACTERISTICS:
Groups:
- Observational Arm: 1. Non-female patients undergoing coronary CTA; 2. Patients undergoing nuclear cardiology stress testing; 3. Patients undergoing invasive coronary angiography.
- Total: Total of all reporting groups
Arm/Group | CCTA Breast Shields | CCTA No Breast Shields | Observational Arm | Total
Number analyzed (Participants) | 50 | 51 | 127 | 228
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (14) | 51 (14) | 51 (12) | 52 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 51 | 92 | 193
  Male | 0 | 0 | 35 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7 | 14
  Not Hispanic or Latino | 46 | 48 | 115 | 209
  Unknown or Not Reported | 0 | 0 | 5 | 5
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 27.6 (6.3) | 28.1 (4.5) | 27.3 (5) | 27.9 (5.5)
Chest circumference (cm) [Mean (Standard Deviation); unit: cm] | 97.6 (11.7) | 97.8 (10.5) | 97.7 (11) | 97.7 (11.1)
Current smokers [Count of Participants; unit: Participants] | 5 | 7 | 15 | 27
Heart rate (beats/min) [Mean (Standard Deviation); unit: beats/min] | 55.2 (5.6) | 56.2 (7.4) | 64 (9) | 55.7 (6.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Excess Double-strand DNA Break Foci Per Cell in Peripheral Blood Samples Post-imaging
Description: The amount of excess DNA double-strand break foci per cell after cardiac computed tomographic angiography (CCTA) in female patients with and without breast shields, minus the amount of foci prior to CCTA. In addition, changes in DNA double-strand breaks from baseline following cardiac testing in the observational arm is being assessed in an observational manner.
Time Frame: Change from baseline double strand DNA breaks at 30 minutes post-imaging
Population: Female patients 18 years or older who were clinically referred to undergo coronary CT angiography between August 2012 and July 2014 at Walter Reed National Military Medical Center (Bethesda, Maryland) were eligible for enrollment.
Measure: Mean (Standard Deviation); unit: gamma-H2AX foci in blood lymphocytes
Groups:
- No Breast Shields; Breast Shields: Within female subset, randomization to wearing bismuth breast shield or not wearing bismuth breast shield (standard of care).
  CCTA: Breast shield placement (randomized) among women.
Arm/Group | No Breast Shields | Breast Shields
Number analyzed (Participants) | 49 | 44
gamma-H2AX foci in blood lymphocytes | 0.183 (0.114) | 0.159 (0.139)
Statistical Analysis 1: Comparison: Breast Shields; Test type: Superiority; p < 0.05, Regression, Linear; Slope = 0.08

ADVERSE EVENTS:
Time Frame: 30 months
Groups:
- CCTA No Breast Shields: Within female subset, randomization to not wearing bismuth breast shield (standard of care).
  .
- Observational Arm: Observational evaluating the dose-related impact of radiation exposure from multiple sources and types on changes in double-stranded DNA breaks.
Arm/Group | CCTA Breast Shields | CCTA No Breast Shields | Observational Arm
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/51 | 0/127
Other Adverse Events (participants affected / at risk) | 0/50 | 0/51 | 0/127

LIMITATIONS AND CAVEATS:
Participants were enrolled at one center and using one CT scanner, variable shield types and shield sizes were not studied, and further work is needed to examine tissue-specific responses to radiation and shielding.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No